CLINICAL TRIAL: NCT04247035
Title: Non-Interventional, Multi-center Registry of Recording of Treatment Standards and Outcomes of Patients With ER/PR Positive, HER2-negative Metastatic Breast Cancer
Brief Title: Τreatment Standards and Outcomes of Patients With ER/PR Positive, HER2-negative Metastatic Breast Cancer
Acronym: MBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic Society of Medical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: Metastatic Breast Cancer
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
• To capture the treatment patterns and clinical characteristics of patients with ER/PR positive, HER2-negative MBC in Greece

DETAILED DESCRIPTION:
* To capture the treatment patterns and clinical characteristics of patients with ER/PR positive, HER2-negative MBC in Greece
* To evaluate the outcome of patients per treatment line (objective response, progression free survival, time to disease progression per line of therapy), overall survival
* To record adverse events per line of therapy
* To recording of the causes of treatment discontinuation per line of therapy

ELIGIBILITY:
Inclusion Criteria:

* Women with histological confirmed ER/PR positive, HER2-negative MBC
* Age >18 years old
* Patients initiating first or second line therapy for ER/PR positive, HER2-negative MBC
* Adequate hematologic, renal and hepatic function
* Signed informed consent (ICF)

Exclusion Criteria:

* Active malignancy other than MBC
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with histological confirmed ER/PR positive, HER2-negative MBC
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-31 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the outcome per treatment line | 5 years
  To evaluate the outcome of patients per treatment line (objective response, progression free survival, time to disease progression per line of therapy), overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Boukovinas, Dr /Phd, Principal Investigator — HeSMO
Locations (1):
- Hellenic Society of Medical Oncology, Athens, Greece